CLINICAL TRIAL: NCT05696691
Title: A Randomized Pilot Trial of Intramuscular Ketamine and Crisis Response Planning for Suicide Prevention in the Emergency Department
Brief Title: Ketamine & Crisis Response Plan for Suicidal Ideation in the ED
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HSC20220426H; UL1TR002645 (NIH)
Record Dates: First submitted 2023-01-12; First posted 2023-01-25 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Suicide
Keywords: Ketamine; Crisis Response Plan; Suicidal Ideation; Emergency Department; Acute Suicidality; Intramuscular Ketamine; Emergency Room
MeSH Terms: conditions — Suicide; Suicidal Ideation; Emergencies | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine and Crisis Response Plan (CRP) (Experimental): Individuals randomized to the experimental arm will receive 100mg intramuscular ketamine injection before completing the Crisis Response Plan. The average timeframe for the experimental arm is anticipated to be approximately 60 minutes of active treatment. Following ketamine administration, the subject will be monitored for 45 minutes with pulse oximetry and recurrent vital signs. The study team will record when the CRP is completed in relation to the ketamine injection.
  Interventions: Drug: Ketamine Hydrochloride; Behavioral: Crisis Response Plan
- Treatment as Usual (No Intervention): Individuals randomized to the no intervention arm will receive routine care from emergency providers and psychiatry staff.

INTERVENTIONS:
Drug: Ketamine Hydrochloride — 100mg IM ketamine to be administered in conjunction with CRP. The ketamine injection will be administered first. Participants will be observed and have vital signs monitored for the first 45 minutes after administering medication in the ED, observing for immediate reactions. Afterwards, participants will continue to be monitored for potential late-term side effects on the inpatient unit. Ketamine will be given only after initial standard of care (SOC) treatment and screening studies have been initiated.
  Other Names: Ketamine
  Arms: Ketamine and Crisis Response Plan (CRP)
Behavioral: Crisis Response Plan — Crisis Response Plan is a brief, empirically-validated, Cognitive-Behavioral Therapy-based one-time therapy, and its administration typically takes 30-60 minutes. It begins with a narrative assessment (allowing patients to "tell their story") and concludes with collaboratively constructed plan that outlines strategies for the patient's self-management of future acute suicidal crises. Patients who engage in CRP are given an index card to keep with them that summarizes the emotional management strategies that they collaboratively generate with the CRP provider.
  Other Names: CRP
  Arms: Ketamine and Crisis Response Plan (CRP)

SUMMARY:
The goal of this randomized pilot trial is to assess the feasibility of administering a combination of 100mg intramuscular (IM) ketamine and Crisis Response Plan (a short psychosocial intervention) for patients with acute suicidality in the context of the Emergency Department setting. This study will assess a combination of a pharmacologic intervention and a psychosocial one. The pharmacologic intervention is a one-time dose of 100mg ketamine delivered intramuscularly (IM) while the patient is in the ED. The psychosocial intervention under study is a brief, patient-centered therapy which takes, on average, 30 minutes to administer. Both interventions will be administered only once. The main questions this study aims to answer are:

* Determine if 100mg of IM ketamine and Crisis Response Plan in combination results in greater short-term reductions in suicidal ideation in adult patients who report acutely elevated suicide risk during an ED visit.
* Examine potential weight-based dose response differences in the reductions in suicidal ideation to determine if future treatment protocols with IM ketamine may benefit from weight-based dosing.

DETAILED DESCRIPTION:
This study is a phase II/III Clinical Pilot Trial. The study participants will be randomized to one of two groups: IM ketamine plus Crisis Response Planning (intervention group) or usual care (control group). Prior to treatment, we will obtain demographic and contact information for patients and for a friend/family member as a collateral reporter of symptom change and safety. As part of informed consent, participants will be warned about the potential for temporary effects of ketamine and provided an enrollment card to inform other care providers of their participation in a ketamine study. Participants will be weighed and complete a series of brief survey assessments. Clinical assessments such as history, physical examination, and routine laboratory testing will be collected as part of usual care. Ketamine and Crisis Response Planning will be administered, and study assessments will be repeated at 120 minutes posttreatment. To ensure the highest level of patient safety, we are proposing only to include patients who have already been cleared for a psychiatric hospitalization. This will also allow for close monitoring of symptom changes during the initial hours and days following treatment. Outcome measures will be collected at two hours, 3 days, and 1 month after the intervention. Research staff will collect assessments by telephone interview and/or visits. Consistent with established protocols, staff will be trained and supervised by STRONG STAR mental health professionals with expertise in evidence-based processes for assessing and responding to suicide risk. Trained and experienced therapists are available to meet with participants to develop a Crisis Response Plan at University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women between the ages of 18 and 70 presenting to the Emergency Department with acute suicidal ideation.
* Patient cleared for admission to the University Hospital inpatient psychiatric unit.
* Decision to admit the patient to the inpatient unit or psychiatric stabilization unit made prior to consent to prevent study procedures from complicating or influencing the disposition and treatment as usual for suicidal patients reporting to the ED.
* Individuals presenting to the ED for other complaints but found to have suicidal ideation necessitating admission will also be eligible.
* Able to read and write English.

Exclusion Criteria:

* Serious mental illness with active and significant signs of psychosis, mania, hallucinations, paranoia, agitation, and drug-induced or other toxidromic symptoms.
* Acute intoxication with clinically significant symptoms (as defined by the attending clinician's assessment of patients' clinical sobriety).
* The patient is not capable of understanding the research procedures and providing informed consent for themselves.
* Lack of reliable means to be available for follow-up assessments (e.g, working mobile phone).
* Persistent resting blood pressure lower than 90/60 or higher than 180/110, or persistent resting heart rate lower than 45 beats/minute or higher than 120 beats/minute.
* Injuries requiring procedural sedation.
* Pregnancy or breast feeding.
* Known hypersensitivity to ketamine.
* Legal or illegal use of ketamine in the previous 90 days.
* End-stage or severe cardiovascular (e.g., ACS or decompensated heart failure), liver, or kidney disease.
* Patient is a prisoner.
* Patient is physically restrained or actively under custody of law enforcement. Once a patient is no longer under custody of law enforcement or physically restrained, the patient may be considered eligible and may consent to voluntary enrollment in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-01-06 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of study interventions | 30 days
  Number of enrolled subjects completing treatment within study parameters, with safety and side-effect profiles at or lower than published rates.

SECONDARY OUTCOMES:
Change in Beck Scale for Suicidal Ideation (SSI) Score | Baseline to 30 days
  The Beck Scale for Suicidal Ideation (SSI) is a 21-item measurement that evaluates the presence and intensity of suicidal thoughts. Each item is scored on a scale from 0-2 with a total score of 0-38; with higher scores indicating higher levels of suicidal ideation.
Change in Depressive Symptoms Index-Suicidality Subscale (DSI-SS) Score | Baseline to 30 days
  The Depressive Symptoms Index-Suicidality Subscale (DSI-SS) is a 4-item measure of suicidal ideation. Respondents rate each item on a 4-point scale ranging from 0-3. Responses are summed, and higher scores reflect more severe suicidal ideation (range: 0-12).
Change in Suicide Visual Analog Scale (S-VAS) Score | Baseline to 30 days
  The Suicide Visual Analog Scale is a 1-item momentary assessment to evaluate severity of suicidal ideation. The item is scored from 0-100 and the total possible score range for the scale is therefore also 0-100. Lower scores indicate less extreme current urges toward self harm, whereas higher scores are indicative of more severe urges.

CONTACTS AND LOCATIONS:
Overall Officials: Robert De Lorenzo, MD, MSM, Principal Investigator — UT Health San Antonio; Romeo Fairley, MD, MPH, Study Director — UT Health San Antonio; Alan Peterson, PhD, ABPP, Study Director — UT Health San Antonio; Stacey Young-McCaughan, RN, PhD, Study Director — UT Health San Antonio
Locations (1):
- University Hospital, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected de-identified participant data that underlie results in a publication will be shared in a peer-reviewed scientific publication once data analysis is complete.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available upon conclusion of the study and dissemination of findings. It will be made available for five (5) years after the conclusion of the study.
Access Criteria: Links to study documents and data will be shared on website following publication of study results to enable the creation and refinement of related projects' study design and procedures.